CLINICAL TRIAL: NCT05671965
Title: Effects of Oral Xylitol on Subsequent Energy Intake, Gastrointestinal Hormones, Glycemic Control, Appetite-related Sensations, and Gastrointestinal Tolerance
Brief Title: Effects of Oral Xylitol on Subsequent Energy Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: PFI-X
Record Dates: First submitted 2022-12-20; First posted 2023-01-05 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Energy Intake; Gastrointestinal Hormones; Glycemic Control; Appetite; Satiation
MeSH Terms: interventions — Xylitol; Sucrose; acetosulfame; Water

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Xylitol (Active Comparator): 20 volunteers receive 33.5g xylitol dissolved in 300mL tap water as an oral pre-load.
  Interventions: Dietary Supplement: Xylitol
- Sucrose (Active Comparator): 20 volunteers receive 33.5g sucrose dissolved in 300mL tap water as an oral pre-load.
  Interventions: Dietary Supplement: Sucrose
- Acesulfame Potassium (Active Comparator): 20 volunteers receive 0.1675g Ace-K dissolved in 300mL tap water as an oral pre-load.
  Interventions: Dietary Supplement: Acesulfame Potassium
- Water (Placebo Comparator): 20 volunteers receive 300mL tap water as an oral pre-load.
  Interventions: Dietary Supplement: Water

INTERVENTIONS:
Dietary Supplement: Xylitol — 33.5g xylitol dissolved in 300mL tap water.
  Other Names: E967-Xylitol
  Arms: Xylitol
Dietary Supplement: Sucrose — 33.5g sucrose dissolved in 300mL tap water.
  Other Names: Saccharose
  Arms: Sucrose
Dietary Supplement: Acesulfame Potassium — 0.1675g Ace-K dissolved in 300mL tap water.
  Other Names: E950-Ace-K
  Arms: Acesulfame Potassium
Dietary Supplement: Water — 300mL tap water.
  Arms: Water

SUMMARY:
The aim of this project is to investigate the effect of xylitol (given as pre-load), compared to sucrose, Ace-K, and water on energy intake during a subsequent ad libitum test meal in healthy participants.

Furthermore, the release of GI hormones, glycemic control, appetite-related sensations, GI tolerance, sweetness and liking in response to the pre-loads will be investigated.

DETAILED DESCRIPTION:
The subjects will participate in four study days. The screening will last 60 minutes, the study days about 4.5 hours each. After a simple-carbohydrate standard dinner, the subjects have to do an overnight fast until the next morning. Subjects will receive fixed equisweet doses of sucrose (33.5g), xylitol (33.5g), Ace-K (0.1675g), or water as oral pre-loads in a blinded, randomized (counterbalanced) fashion (t = -15 min). Fifteen minutes after the administration (t = 0 min), a standard solid test meal will be presented and ad libitum energy intake will be measured. The end of the test meal will be after 20 minutes or as soon as the subject stops eating for more than 5 minutes. Blood samples (to measure: glycemic control and GI hormones) will be collected at t = -16, t = -1, t = 15, t = 30, t = 60, t = 90, t = 120, t = 150, t = 180 min and appetite-related sensation rating will be collected at t = -16, t = -1, t = 15, t = 30, t = 60, t = 90, t = 120, t = 150, t = 180 min. GI symptoms and nausea are assessed at t = -16, -1, 30, 60, 120 and 180 min. At t = -10 min subjects are asked to rate the perceived sweetness and liking of the pre-load and at t = 180 min the perceived liking of the test meal.

ELIGIBILITY:
Inclusion Criteria:

* Healthy normal weight participants (10 male and 10 female) with a body-mass index (BMI) of 19.0-24.9 kg/m2
* Age 18-55 years
* Stable body weight (± 5%) for at least three months
* Able to give informed consent as documented by signature

Exclusion Criteria:

* Fructose intolerance
* Pre-existing diet (vegetarian, vegan, sugar free, no breakfast)
* Pre-existing regular consumption of xylitol and/or Ace-K (> 1/week)
* Chronic or clinically relevant acute infections/diseases
* Regular intake of medications, except contraceptives
* Pregnancy: although no contraindication, pregnancy might influence metabolic state.
* Substance abuse (more than 1 glass wine/beer per day; consumption of cannabis, cocaine, heroin, etc.)
* Shift worker
* Participation in another study with investigational drug within the 30 days preceding and during the present study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2023-01-27 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
Effect of xylitol on energy intake during a subsequent ad libitum test meal | Total energy intake will be measured from t = 0 until t = 20 minutes or as soon as the as the subject stops eating for more than 5 minutes.
  Fifteen minutes after the administration of the pre-loads (t = 0 minutes), a standard solid test meal will be presented and ad libitum energy intake will be measured.

SECONDARY OUTCOMES:
Effects on GI hormone response - GLP-1 | Blood will be drawn at the following time points :t = -16, t = -1 (before the administration of the pre-load), t = 15, t = 30, t = 60, t = 90, t = 120, t = 150, t = 180 minutes (after the administration of the pre-load).
  GLP-1 will be quantified using a non-radioactive highly sensitive sandwich ELISA (MSD V-PLEX - #K1503PD) in the presence of a chemiluminescent substrate.
Effects on GI hormone response - PYY | Blood will be drawn at the following time points :t = -16, t = -1 (before the administration of the pre-load), t = 15, t = 30, t = 60, t = 90, t = 120, t = 150, t = 180 minutes (after the administration of the pre-load).
  PYY-3-36 will be quantified using a non-radioactive high sensitive sandwich ELISA (Millipore - # EZHPYYT66K).
Effects on GI hormone response - CCK | Blood will be drawn at the following time points: t = -16, t = -1 (before the administration of the pre-load), t = 15, t = 30, t = 60, t = 90, t = 120, t = 150, t = 180 minutes (after the administration of the pre-load).
  Plasma cholecystokinin (CCK) levels will be measured with a sensitive radioimmunoassay using a highly specific antiserum (No. 92128)
Effects on GI hormone response - ghrelin | Blood will be drawn at the following time points: t = -16, t = -1 (before the administration of the pre-load), t = 15, t = 30, t = 60, t = 90, t = 120, t = 150, t = 180 minutes (after the administration of the pre-load).
  Octanoylated ghrelin will be measured by a radioimmunoassay with 125I [Tyr24] human ghrelin [1-23] as tracer and a rabbit antibody against human ghrelin [1-8] (final dilution 1/100000), which does not cross-react with desoctanoylated ghrelin.
Effects on glycemic control - plasma glucose | Blood will be drawn at the following time points: t = -16, t = -1 (before administration of the pre-load), t = 15, t = 30, t = 60, t = 90, t = 120, t = 150, t = 180 minutes (after the administration of the pre-load).
  Glucose will be measured by a glucose oxidase method (Rothen Medizinische Laboratorien AG, Basel, Switzerland).
Effects on glycemic control - plasma insulin | Blood will be drawn at the following time points: t = -16, t = -1 (before the administration of the pre-load), t = 15, t = 30, t = 60, t = 90, t = 120, t = 150, t = 180 minutes (after the administration of the pre-load).
  Insulin will be quantified using a chemiluminescent microparticle immunoassay (chemiflex) reagent kit (#8k41; Abbott) and the relative light units detected by the ARCHITECT optical system (model: CI4100; Abbott).
Effects on glycemic control - plasma c-peptide | Blood will be drawn at the following time points: t = -16, t = -1 (before administration of the pre-load), t = 15, t = 30, t = 60, t = 90, t = 120, t = 150, t = 180 minutes (after the administration of the pre-load).
  C-peptide will be measured with a commercially available sandwich ELISA kit from Millipore (Millipore - # EZHCP-20K).
Effects on glycemic control - plasma glucagon | Blood will be drawn at the following time points: t = -16, t = -1 (before the administration of the pre-load), t = 15, t = 30, t = 60, t = 90, t = 120, t = 150, t = 180 minutes (after the administration of the pre-load).
  Glucagon concentrations in plasma will be measured after extraction of plasma with 70% ethanol (vol/vol, final concentration). The antibody is directed against the C-terminus of the glucagon molecule (antibody code no. 4305) and therefore mainly measures glucagon of pancreatic origin.
Effects on appetite-related sensations | Visual analogue scales will be recorded at the following time points: t = -16, t = -1 (before the administration of the pre-loads), t = 15, t = 30, t = 60, t = 90, t = 120, t = 150, t = 180 minutes (after the administration of the pre-loads).
  Appetite perceptions (feelings of: a) hunger, b) satiety) are assessed by visual analogue scale (VAS). Visual analogue scales consist of a horizontal, unstructured, 10-cm line representing the minimum (0.0 points) to the maximum rating (10.0 points). Subjects assign a vertical mark across the line to indicate the magnitude of their subjective sensation at the present time point. The measurement is quantified by the distance from the left end of the line (minimum rating) to the subject's vertical mark.
Effects on GI tolerance | GI tolerance will be recorded at t = -16, -1 (before the administration of the pre-load), 30, 60, 120 and 180 minutes (after the administration of the pre-load).
  GI symptoms will be assessed by use of a checklist including the following questions: abdominal pain, nausea, vomiting, diarrhea, borborygmic, abdominal distension, eructation and increased flatus.
Sweetness of pre-load | Sweetness of the pre-load will be recorded at t = -10 minutes.
  Sweetness is assessed by gLMS. General Labeled Magnitude Scales consist of an unequal, vertical line, which is marked with quasi-logarithmic verbal anchors describing different intensities (e.g. "strongest imaginable", "barely detectable"). Participants are instructed to place a mark on the line where their perceived intensity of sensation lies.
Liking ot the pre-load | Liking of the pre-load will be recorded at t = -10 minutes.
  Liking is assessed by gLMS. General Labeled Magnitude Scales consist of an unequal, vertical line, which is marked with quasi-logarithmic verbal anchors describing different intensities (e.g. "strongest imaginable", "barely detectable"). Participants are instructed to place a mark on the line where their perceived intensity of sensation lies.
Liking of the test meal | Liking of the test meal will be recorded at t = 180 minutes.
  Liking is assessed by gLMS. General Labeled Magnitude Scales consist of an unequal, vertical line, which is marked with quasi-logarithmic verbal anchors describing different intensities (e.g. "strongest imaginable", "barely detectable"). Participants are instructed to place a mark on the line where their perceived intensity of sensation lies.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Christin Meyer-Gerspach, Principal Investigator — St. Clara Research Ltd.
Locations (1):
- St. Claraspital, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Flad E, Altstadt A, Beglinger C, Rehfeld JF, Van Oudenhove L, Wolnerhanssen BK, Meyer-Gerspach AC. Effects of Oral Xylitol, Sucrose, and Acesulfame Potassium on Total Energy Intake During a Subsequent ad libitum Test Meal: A Randomized, Controlled, Crossover Trial in Healthy Humans. Nutrients. 2025 Jan 29;17(3):484. doi: 10.3390/nu17030484. PMID 39940340